CLINICAL TRIAL: NCT04999943
Title: A Randomized, Open-label, Clinical Trial to Compare the Safety and Efficacy of Hypomemylating Agents Monotherapy and Combination With eDC Therapy for Elderly Patients With Myelodysplastic Syndrome
Brief Title: Hypomemylating Agents Combination With eDC Therapy for Elderly Patients With Myelodysplastic Syndrome
Acronym: eDC-MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2107-Hem-1-eDC
Record Dates: First submitted 2021-06-30; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Myelodysplastic Syndromes; Dendritic Cell; Hypomethylating Agents; Immunotherapy
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypomemylating agent monotherapy (Active Comparator): Azacitidine 100mg/ times. d × for 10 days (28 days for one cycle) or Decitabine 25mg/ times. d × 5 days ( 28 days is one cycle)
  Interventions: Biological: DC vaccine
- Combined cellular immunotherapy（eDC）with Hypomemylating agent therapy (Experimental): Azacitidine 100mg/ times. d × for 10 days (28 days for one cycle) or Decitabine 25mg/ times. d × 5 days ( 28 days is one cycle) with Dendritic Cell (DC) Vaccination Expressing WT1/hTERT/Survivin
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — EDC cell therapy collection and administration process. Collection of PBMC for preparation of DC cells for patients with autologous DC cells, patient PBMC was collected 10-16 weeks before administration for the preparation and large-scale culture of DC cells. For the patients with matched DC cells, a small amount of peripheral blood was taken for HLA typing 4 weeks before administration, and then the matched DC cells were cultured on a large scale.

SUMMARY:
The purpose of this study is to optimize the traditional treatment scheme and explore the cure scheme for the elderly by combining the existing mature treatment technology. The primary aim of this innovative immunotherapy using WT1/hTERT/Survivin-loaded DCs is to determine whether this novel DC vaccination is safe and can significantly prevent clinical relapse and increase survival of MDS patients.

DETAILED DESCRIPTION:
Objective Myelodysplastic syndrome (Myelodysplasticsyndromes,MDS) is a highly age-related malignant clonal disease of the hematological system, which is characterized by pancytopenia and transformation to leukemia. In China, the median age of onset of MDS is 70 years old, and the incidence increases with age. It is the most common malignant tumor in the elderly, which seriously threatens the health and survival of the elderly. The 3-year survival rate of traditional combination chemotherapy or demethylation therapy is less than 20%.

ELIGIBILITY:
Inclusion Criteria:

1. elderly MDS patients;
2. aged more than 60 years old, general condition, ECOG score less than 1;
3. normal function of heart, liver and kidney, serum bilirubin ≤ 35 umol / L; serum creatinine ≤ 150 umol / L;
4. patients are unsuitable or unwilling to receive hematopoietic stem cell transplantation;
5. subjects sign informed consent.

Exclusion criteria:

1. serious infection was not controlled before treatment;
2. contraindications for the use of dexitabine and azacytidine;
3. other cases that did not meet the admission criteria.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
OS | at study completion, an average of 3 years
  Overall survival

SECONDARY OUTCOMES:
the Incidence of Treatment Adverse Events | at study completion, an average of 3 years
  The primary objective of this single-arm phase I clinical study is to determine the Incidence of Treatment Adverse Events in elder MDS or MDS/AML patients.
RR | at study completion, an average of 3 years
  Relapse rate
RFS | at study completion, an average of 3 years
  Relapse-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Liangding Hu, Prof., Study Chair — the Fifth Medical Center the PLA General Hospital
Locations (1):
- Department of hematology, Beijing, China